CLINICAL TRIAL: NCT01262690
Title: A Phase 1 Ascending Single Dose Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-05230901 Administered Subcutaneously To Healthy Subjects
Brief Title: A Study In Healthy Subjects Of Single Doses of PF-05230901 Injected Under The Skin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on 21-Sept-2011 due to the emergent safety concern of sensory symptoms.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B2291001; TAM-163 FIH Study; 3279K1-1000
Record Dates: First submitted 2010-11-23; First posted 2010-12-17 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cachexia
Keywords: First-in-human (FIH); Single Ascending Dose (SAD) Study; TAM-163; PF-05230901; Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose (Experimental): 6 treated, 3 placebos
  Interventions: Drug: PF-05230901

INTERVENTIONS:
Drug: PF-05230901 — Single ascending doses of PF-05230901 in separate cohorts of subjects; each cohort consists of 6 subjects treated with PF-05230901 and 3 subjects treated with placebo.
  Other Names: TAM-153
Drug: PF-05230901 — Single dose SC
  Other Names: TAM-163

SUMMARY:
This study will examine whether a single dose of PF-05230901 is safe and well tolerated when given to healthy volunteers by injection under the skin. An additional objective is to measure the blood concentrations of PF-05230901. Each dose will be tested in a different group of subjects starting from the lowest dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* History of seizures, including childhood seizures.
* History of movement disorders or related neurological conditions.
* History of head trauma associated with loss of consciousness.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | 35 days
Incidence and severity of clinical laboratory abnormalities. | 35 days
Mean change from baseline in vital signs. | 35 days
Mean change from baseline in 12-lead electrocardiogram (ECG) parameters. | 35 days
Incidence and severity of findings during the neurological examination. | 35 days

SECONDARY OUTCOMES:
Plasma concentrations | 14 days
Anti-drug antibodies | 35 days
Appetite and food consumption | 13 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2291001&StudyName=A%20Study%20In%20Healthy%20Subjects%20Of%20Single%20Doses%20of%20PF-05230901%20Injected%20Under%20The%20Skin